CLINICAL TRIAL: NCT02139267
Title: A Randomized, Open-label, Multi-center, Phase 2 Clinical Trial to Determine the Optimal Dose and Evaluate the Safety of GX-188E, a DNA-based Therapeutic Vaccine, Administered Intramuscularly by Electroporation (EP) in HPV Type 16 and/or 18 Positive Patients With Cervical Intraepithelial Neoplasia 3 (CIN 3)
Brief Title: Dose-finding, Safety Study of Plasmid DNA Therapeutic Vaccine to Treat Cervical Intraepithelial Neoplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GX-188E_CIN3_P2
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: CIN3; Cervical Intraepithelial Neoplasia; High-Risk HPV; HPV Infection; Neoplasm; Precancerous Diseases; Uterine Diseases; Genital Diseases, Female
MeSH Terms: conditions — Uterine Cervical Dysplasia; Papillomavirus Infections; Neoplasms; Uterine Diseases; Genital Diseases, Female | interventions — GX-188 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1mg of GX-188E per dose (Experimental): 1mg of GX-188E per dose will be administered on 1mg group participants through intramuscular route using EP device. The injection points are at 0 week, 4 week and 12 week.
  Interventions: Biological: GX-188E
- 4mg of GX-188E per dose (Experimental): 4mg of GX-188E per dose will be administered on 4mg group participants through intramuscular route using EP device. The injection points are at 0 week, 4 week and 12week.
  Interventions: Biological: GX-188E

INTERVENTIONS:
Biological: GX-188E — DNA vaccine administered via IM route using TDS-IM electroporation device
  Other Names: DNA therapeutic vaccine

SUMMARY:
The purpose of this study is to determine the optimal dose of GX-188E for the Phase 3 and access the efficacy and safety of GX-188E according the protocol in patients with Cervical Intraepithelial Neoplasia 3 (CIN3).

DETAILED DESCRIPTION:
Subjects who are eligible for this study are allocated to one of the two treatment groups of GX-188E. All Subject received GX-188E intramuscularly using the electroporator(EP) on alternating deltoid muscles which will be performed totally three times during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed informed consent form after receiving education about this study and the investigational product.
2. Female aged between 19 and 50 years
3. Positive test results for HPV Type 16 and/or Type 18
4. Histopathologically-confirmed Cervical Intraepithelial Neoplasia 3
5. Entire cervical area including entire squamocolumnar junction is visualized through colposcopy
6. Eligible based on screening test results.
7. Promised not to get pregnant throughout the study

Exclusion Criteria:

1. Suspected Adenocarcinoma in situ
2. Malignant cancer more than Stage I
3. Pregnancy or breastfeeding
4. Participation in clinical trials within 30 days of the screening visit
5. Administration of immunosuppressant or immunomodulator within 6 months prior to the enrolment
6. Administered with systemic steroid(as a standard with Prednisolone, more than 20mg/day for every 14 days or more) within 3 months of Day 1(including ointment, eye drops, inhalated or nasal, intra-ligamental or intra-articular injection, but not applicable if injected every other day
7. Administered any blood products within 3 months prior to the screening visit
8. Administered any vaccine within 4 weeks prior to the screening visit(ex. Hepatitis A, Hepatitis B, Influenza, Td etc.)
9. Positive serum test results for hepatitis C virus, hepatitis B virus surface antigen(HBsAg) or HIV
10. Severe hepatopathy which is Class C according to Child-Pough's classification
11. Severe renal dysfunction where the creatinine clearance(CLcr) is lower than 30ml/min
12. CPK test results more than 2.5 times the upper limit of normal
13. Predisposed to inflammatory reaction due to use of medical devices such as electroporation within 30 days of screening visit
14. History of severe adverse drug events or severe allergic diseases
15. History of epilepsy or convulsion within 2 years prior to the screening visit
16. At the discretion of the investigator, the skin condition covering deltoid muscles, within 2cm of the intended sites of injection, is not suitable for injection due to infection, ulcer, edema, tattoo, scar, injury etc.
17. The thickness of skin fold covering deltoid muscles, intended injection sites, > 40mm
18. Any orthopedic artificial implant around the intended sites of electroporation (deltoid muscles)
19. Sinus bradycardia whose resting heart rate < 50 beats/min
20. Pre-excitation syndrome such as Wolff-Parkinson-White syndrome
21. Abnormal electrocardiography(ECG) including arrhythmia
22. Artificial implants or metallic implants
23. Any other ineligible condition at the discretion of the investigator that would be ineligible to participate the study

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The Rate of Participants with Histopathological Regression of Cervical Lesions to CIN1 or Less | 20 weeks

SECONDARY OUTCOMES:
The Rate of Participants Whose Result Inverted Negative in HPV DNA test | 20 weeks
The rate of HPV E6, E7-specific ELISPOT responder defined in the protocol | 20 weeks
Cytological Changes of the Cervical Lesions | 20 weeks
The Rate of Adverse Events and the Related Features after Administration of Investigational Product | 20 weeks
The Rate of Solicited Adverse Events and the Related Features | 20 weeks
Data in Physical examination, Vital signs, Electrocardiography, Clinical Laboratory Test Results Related to Investigational Product | 20 weeks
Mean Value of Visual Analogue Scale on Pain Intensity | 20 weeks
Flt-3L Serum Concentration | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Park Jong-Sup, M.D., Principal Investigator — The Catholic University of Korea; Kim Tae-Jin, M.D., Principal Investigator — Cheil General Hospital & Women's Healthcare Center; Lee Jae-kwan, M.D., Principal Investigator — Korea University Guro Hospital; Cho Chi-heum, M.D., Principal Investigator — Keimyung University Dongsan Medical Center
Locations (4):
- South Korea (4):
  - Keimyung University Dongsan Medical Center, Daegu
  - Cheil General Hospital & Women's Healthcare Center, Seoul
  - The Catholic University of Korea Seoul St.Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul

REFERENCES:
- [Derived] Cho HW, Jeong S, Song SH, Kim YT, Kim JW, Cho CH, Hur SY, Chang SJ, Kim YM, Lee JK. A phase 1/2a, dose-escalation, safety, and preliminary efficacy study of the RKP00156 vaginal tablet in healthy women and patients with cervical intraepithelial neoplasia 2. J Gynecol Oncol. 2024 Jul;35(4):e52. doi: 10.3802/jgo.2024.35.e52. Epub 2024 Jan 24. PMID 38330377